CLINICAL TRIAL: NCT03995537
Title: Monocytic Expression of HLA-DR After Liver Transplantation
Acronym: EdMonHG
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0116; 2019-A00954-53 (Other: ID-RCB)
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Liver Diseases; Liver Transplantation; Cirrhosis, Liver
Keywords: liver transplantation; Liver Diseases
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — One samples of Ethylenediaminetetraacetic acid (EDTA) (4 millilitre (mL)), one Heparin sample (4mL) and one PAXgene® sample (2.5mL) will be collected:
  * at inclusion
  * between inclusion and LT in case of major clinical change
  * During the pre-transplant follow-up 3 months after inclusion, for patients who have not been transplanted within 3 months following inclusion. At 6 months post-inclusion, non-transplanted patients will terminate the study prematurely
  * at day 1 after LT
  * 2 times a week after the LT for a maximum of 1 month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with severe liver disease waiting liver transplant: Only patients with the most frequent LT indications will be eligible: complicated cirrhosis of hepatocellular carcinoma (HCC), acute or chronic decompensation of cirrhosis, with or without multi-visceral failure and fulminant hepatitis.
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — Samples will be collected at the inclusion and repeated if necessary before LT, including one 4 mL EDTA sample and one 4 mL Heparin sample and one 2.5 mL PAXgene® sample, allowing the HLA-DR assay to be performed with also plasma aliquots and messenger RNAs.
  Same samples will also be collected :
  * between inclusion and LT in case of major clinical change
  * During the pre-transplant follow-up 3 months after inclusion, for patients who have not been transplanted within 3 months after inclusion
  * at day 1 after LT
  * 2 times a week after the LT for a maximum of 1 month
  Biological data will be collected at those different times.

SUMMARY:
A defect of the immune response has been described in patients with severe liver disease. This immune-paresis is partly driven by a compensatory anti-inflammatory response following a systemic inflammatory response syndrome and affects the innate immune response. The innate immune defect has been described in patients with advanced cirrhosis and more significantly in patients with acute liver failure or acute on chronic liver failure (ACLF). The monocytes/macrophages pro-inflammatory response and finally the antimicrobial response are thus strongly impaired, leading to higher sepsis risk. The monocytes/macrophages phenotype associated with these functional alterations has been widely described, with a weaker expression of Human Leukocyte Antigen - DR isotype (HLA-DR) on the monocytes surface, correlated with poor outcomes. The low monocytic expression of HLA-DR, its functional and clinical impact has been widely described in the context of septic shock with similar pathophysiological mechanisms.

Liver transplantation (LT) is often the only therapeutic option for patients with advanced liver failure. Post-transplant survival of the most severe patients is similar to the survival in the whole population of LT patients, but the complication rate remains higher, with a major risk of infection. Currently used immunosuppression protocols do not take into account the quality of pre-transplant immune response. Some treatments, such as corticosteroids, which are widely used for the induction of post-transplant immunosuppression, may affect the innate immune response. However, it has been shown that low expression of post-transplant monocyte HLA-DR was associated with a greater risk of septic complication.

The general objective of this study is to focus on the evolution of a robust marker of immune dysfunction, HLA-DR monocyte expression, before and following LT, and to analyse its post LT expression depending on the level of pre-transplant expression as well as its association with post-transplant complications. This study will bring new insights for the design of a prospective study on the relevance of adapting post-transplant immunosuppression protocols to HLA-DR expression on monocytes surface, which is a robust marker of the innate immune response.

Evaluation of innate immune dysfunction pre-LT by quantification of monocytic HLA-DR expression and monitoring of its post-LT kinetics may be relevant for assessing post-transplant immune status and adapting immunosuppressive therapy. A descriptive, observational study associating clinical and biological data is needed to confirm the relevance of HLA-DR expression quantification on the surface of monocytes in a population of selected patients, before and after LT. These data will allow setting up a prospective interventional study reporting the possible benefit of post-transplant immunosuppressive treatment modulation, according to the HLA-DR monocyte dosage and its kinetics evolution.

The main objective of this study is to describe the association between evolution of monocytic HLA-DR expression on monocytes/macrophages surface during the first month after LT and the occurrence of one of the 2 following clinical events reflecting a post LT immune dysfunction (acute cell rejection and sepsis).

ELIGIBILITY:
Inclusion Criteria:

* Patients waiting for LT in the LT center of the Groupement Hospitalier Nord, and in the hepato-gastroenterology department of the Groupement hospitalier centre, Hospices Civils de Lyon, presenting :

  * Cirrhosis

    * Complicated with hepatocellular carcinoma
    * Or chronically decompensated (recurrent gastrointestinal bleeding, refractory ascites, portopulmonary or hepatopulmonary syndrome, chronic liver failure)
    * Or with acute decompensation, with or without multi-visceral failure
  * Or fulminant hepatitis
* Patient eligible for the standard immunosuppression protocol (induction with anti-Interleukin-2 (IL2) (Day1 and Day4) and then corticosteroids for a minimum of 7 days associated with tacrolimus and mycophenolate mofetil)
* Patient having theoretical access to LT within <3 months (head of local and / or national waiting list)

Exclusion Criteria:

* Minor or adult patient under tutorship or curatorship
* Pregnant and lactating woman
* Patient without liberty
* Patient not affiliated to social security
* Refusal to participate in the study
* Patient enrolled in "super-emergency" outside working days
* Patients waiting for LT without underlying liver disease (healthy liver HCC, cholangiocarcinoma, primary tumor metastases, amyloidosis, Rendu Osler disease, dominant biliary disease such as recurrent angiocholitis without underlying cirrhosis)
* Patient who already had a LT
* Patient who received a multi-organ transplant (liver + kidney / heart / lung / intestine)
* Patient on immunosuppressive therapy before hepatic transplant (other than corticosteroids)
* Patient not eligible for standard immunosuppression protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe liver disease waiting for LT. Only patients with the most frequent LT indications will be eligible: complicated cirrhosis of hepatocellular carcinoma (HCC), acute or chronic decompensation of cirrhosis, with or without multi-visceral failure and fulminant hepatitis.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
number of receptors expressed by monocytes | 7 months
  Primary outcome will be the kinetics of HLA-DR expression on the monocytes / macrophages surface during the first month after LT as a function of pre-LT status (Nadir, normalization delay of HLA-DR expression) and its association with 2 clinical events reflecting post-LT immune dysfunction (acute cell rejection and sepsis).
  Expression of HLA-DR is measured by the number of receptors expressed by monocytes and measured by flow cytometry at different times: at inclusion (D0), Month 3, Month 6, the day of LT and twice a week for 1 month in post LT.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service d'hépato gastroentérologie hôpital Edouard Herriot Groupement hospitalier centre, Lyon
  - Hopital de la Croix-Rouse, service de réanimation chirurgicale, Lyon
  - Hospital de la Croix Rousse, service d'hépatologie, Lyon

REFERENCES:
- [Derived] Delignette MC, Riff A, Antonini T, Soustre T, Bodinier M, Peronnet E, Venet F, Gossez M, Pantel S, Mabrut JY, Muller X, Mohkam K, Villeret F, Erard D, Dumortier J, Zoulim F, Heyer L, Guichon C, Blet A, Aubrun F, Monneret G, Lebosse F. Individual mHLA-DR trajectories in the ICU as predictors of early infections following liver transplantation: a prospective observational study. Crit Care. 2025 Feb 18;29(1):79. doi: 10.1186/s13054-025-05305-x. PMID 39966934